CLINICAL TRIAL: NCT06629597
Title: A Randomized, Controlled, Multicenter Phase III Clinical Study of YL201 Versus Investigator's Choice of Chemotherapy in Subjects with Recurrent or Metastatic Nasopharyngeal Carcinoma Who Have Failed Prior PD-(L)1 Inhibitor and At Least Two Lines of Chemotherapy
Brief Title: A Phase III Study of YL201 in Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YL201-CN-301-01
Record Dates: First submitted 2024-09-24; First posted 2024-10-08 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- YL201 (Experimental): Participants are randomized to receive YL201 monotherapy intravenously on Day 1 of each 3-week cycle at RP3D dose level, until progressive disease (PD), unacceptable toxicity, or withdrawal of consent as specified in the protocol.
  Interventions: Drug: YL201
- Investigator's choice of chemotherapy, including docetaxel, capecitabine, or gemcitabine (Active Comparator): Participants are randomized to receive docetaxel/capecitabine/gemcitabine every 3 weeks per prescribing information, until PD, unacceptable toxicity, or withdrawal of consent as specified in the protocol.
  Interventions: Drug: Docetaxel; Drug: Capecitabine; Drug: Gemcitabine

INTERVENTIONS:
Drug: YL201 — YL201 will be administered intravenously on Day 1 of each 3-week cycle at RP3D dose level.
  Arms: YL201
Drug: Docetaxel — Docetaxel will be administered intravenously at 75 mg/m2 on Day 1 of each 3-week cycle.
  Arms: Investigator's choice of chemotherapy, including docetaxel, capecitabine, or gemcitabine
Drug: Capecitabine — Capecitabine will be administered orally at 1000 mg/m2 twice a day (BID) on Days 1 to 14 of each 3-week cycle
  Arms: Investigator's choice of chemotherapy, including docetaxel, capecitabine, or gemcitabine
Drug: Gemcitabine — Gemcitabine will be administered intravenously at 1000 mg/m2 on Day 1 and 8 of each 3-week cycle
  Arms: Investigator's choice of chemotherapy, including docetaxel, capecitabine, or gemcitabine

SUMMARY:
This study was designed to compare the efficacy and safety of YL201 with Investigator's choice of chemotherapy in subjects with recurrent or metastatic nasopharyngeal carcinoma who have failed prior PD-(L)1 inhibitor and at least two lines of chemotherapy.

DETAILED DESCRIPTION:
The primary objective of this study is to assess whether treatment with YL201 prolongs overall survival (OS) and increases objective response rate (ORR) by blinded independent central review (BICR) compared with treatment of investigator's choice of chemotherapy among subjects with recurrent or metastatic nasopharyngeal carcinoma.

The secondary objectives of the study are to further evaluate the efficacy, safety, pharmacokinetics, and immunogenicity of YL201, and the correlation between B7-H3 expression level and the efficacy of YL201.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written informed consent form (ICF).
2. Aged ≥18 years and ≤75 years, male or female.
3. ECOG performance status score of 0 or 1.
4. Life expectancy ≥ 3 months.
5. Histologically or cytologically confirmed recurrent or metastatic nasopharyngeal carcinoma that is not amenable to curative treatment.
6. Have failed prior treatment with PD-(L)1 inhibitors and at least two lines of chemotherapy.
7. Suitable for treatment with investigator's choice of chemotherapy (docetaxel, capecitabine, or gemcitabine).
8. At least one measurable lesion according to RECIST v1.1.
9. Subjects are willing to provide the archived or freshly obtained tumor tissue (freshly obtained or archived) for detection of B7-H3 expression
10. Adequate organ function.

Exclusion Criteria:

1. History of other malignant tumors within 5 years prior to the first dose of study drug. Subjects who have been cured of other tumors by local therapy, such as basal cell carcinoma, squamous cell carcinoma of skin, bladder cancer in situ, cervical carcinoma in situ, or breast cancer in situ, are not excluded.
2. Previously received B7-H3-targeted drug therapy, including antibody, antibody-drug conjugate (ADC), and chimeric antigen receptor T cell (CAR-T).
3. Prior treatment with a topoisomerase I inhibitor or an antibody-drug conjugate containing a topoisomerase I inhibitor.
4. Inadequate washout period for prior anti-tumor treatment before the first dose of study drug.
5. Received radical radiotherapy within 4 weeks prior to the first dose of study drug; local palliative radiation for symptom control is allowed, but treatment must be completed at least 2 weeks prior to the first dose of study drug, and there is no plan for additional radiotherapy to the same lesion.
6. Received systemic steroids or other immunosuppressive therapy within 2 weeks before the first dose of study drug.
7. Received any live vaccine within 4 weeks before the first dose of study drug or intend to receive a live vaccine during the study.
8. Presence of brain stem or meningeal metastases, spinal cord metastases or compression.
9. Presence of central nervous system (CNS) metastasis. Participants with treated brain metastases are eligible if the metastases are asymptomatic and stable, and no immediate local or systemic treatment is needed within 2 weeks before the first dose.
10. Has an uncontrolled concurrent disease.
11. Presence of severe uncontrolled cardiovascular disorder.
12. History of interstitial lung disease (ILD) or pneumonitis that required corticosteroids, or current ILD/ pneumonitis.
13. Concomitant pulmonary disorder leading to clinically severe respiratory impairment.
14. Chronic autoimmune or inflammatory diseases requiring systemic therapy within 2 years prior to the first dose or currently receiving systemic therapy.
15. Clinical symptoms of pleural effusion, pericardial effusion, or ascites or requiring relevant repeated drainage.
16. Serious infections within 4 weeks prior to the first dose.
17. Known active pulmonary tuberculosis (TB).
18. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
19. Unresolved toxicities from previous antitumor therapy.
20. Known allergy to any component of the study drug; history of severe allergic reactions or known history of severe hypersensitivity to other monoclonal antibodies or recombinant proteins, or history of severe infusion reactions.
21. Pregnancy, breastfeeding, or women planning to become pregnant or breastfeed during the study.
22. Any illness, medical condition, organ system dysfunction, or social situation deemed by the investigator to be likely to interfere with a subject's ability to sign ICF, adversely affect the subject's ability to cooperate and participate in the study, or compromise the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare the ORR of YL201 versus investigator's choice of chemotherapy in recurrent or metastatic nasopharyngeal carcinoma assessed by BICR based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). | Approximately within 36 months
  ORR is defined as the proportion of subjects who achieve a best overall response (BOR) of complete response (CR) or partial response (PR).
To compare the OS of YL201 versus investigator's choice of chemotherapy in recurrent or metastatic nasopharyngeal carcinoma. | Approximately within 36 months
  OS defined as the time interval from the randomization to death from any cause.

SECONDARY OUTCOMES:
To compare the ORR of YL201 versus investigator's choice of chemotherapy in recurrent or metastatic nasopharyngeal carcinoma assessed by Investigator. | Approximately within 36 months
  ORR is defined as the proportion of subjects who achieve a best overall response (BOR) of complete response (CR) or partial response (PR).
To compare the PFS of YL201 versus investigator's choice of chemotherapy in recurrent or metastatic nasopharyngeal carcinoma assessed by BICR and Investigator. | Approximately within 36 months
  PFS defined as the time interval from randomization to the first documented PD or death due to any cause, whichever occurs first.
To compare the DOR of YL201 versus investigator's choice of chemotherapy in subjects with recurrent or metastatic nasopharyngeal carcinoma assessed by BICR and Investigator. | Approximately within 36 months
  DOR defined as the time interval from the first documentation of response (CR or PR) to the first documentation of PD or death, whichever occurred first.
To compare the DCR of YL201 versus investigator's choice of chemotherapy in subjects with recurrent or metastatic nasopharyngeal carcinoma assessed by BICR and Investigator. | Approximately within 36 months
  DCR is defined as the proportion of subjects with a BOR of CR, PR, or stable disease (SD).
To compare the TTR of YL201 versus investigator's choice of chemotherapy in subjects with recurrent or metastatic nasopharyngeal carcinoma assessed by BICR and Investigator. | Approximately within 36 months
  TTR is defined as the time interval from randomization to the first documentation of response (CR or PR).
Evaluate the incidence and severity of adverse events (AEs) of YL201 | Approximately within 36 months
  AEs are assessed based on NCI CTCAE v5.0.
Characterize the PK parameter AUC | Approximately within 36 months
Characterize the PK parameter Cmax | Approximately within 36 months
Characterize the PK parameter Ctrough | Approximately within 36 months
Characterize the PK parameter CL | Approximately within 36 months
Characterize the PK parameter Vd | Approximately within 36 months
Characterize the PK parameter t1/2 | Approximately within 36 months
Assessment of the number of subjects who are Anti-Drug Antibody (ADA)-positive at any time and who have a treatment-emergent ADA. | Approximately within 36 months
Assessment of B7H3 expression level in tumor tissue and the correlation between the expression level and the efficacy of YL201. | Approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China